CLINICAL TRIAL: NCT06215157
Title: A Comparison of Stroke Volume Variation for Prediction of Fluid Responsiveness Measured by Thoracic Electrical Bioimpedance and FloTrac/Vigileo
Brief Title: A Comparison of Stroke Volume Variation for Prediction of Fluid Responsiveness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TEB-Zhoujie
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Stroke Volume Variation; SVV-FloTrac; Thoracic Electrical Bioimpedance; Fluid Responsiveness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flotrac Group (Active Comparator): In this group,an arterial catheter was inserted preoperatively. An indwelling radial artery catheter was connected to the hemodynamic monitoring system (EV1000; Edward Lifesciences Corp., Irvine, CA, USA) via FloTrac™ (Edwards Lifesciences Corp.) sensors.
  Interventions: Device: Flotrac Group
- BioZ Group (Experimental): In this group,haemodynamic parameters were collected simultaneously by the thoracic bioimpedance (BioZ.com™) monitoring.
  Interventions: Device: BioZ Group

INTERVENTIONS:
Device: Flotrac Group — Haemodynamic parameters were collected simultaneously by the Flotrac monitoring.
  Arms: Flotrac Group
Device: BioZ Group — Haemodynamic parameters were collected simultaneously by the thoracic bioimpedance (BioZ.com™)monitoring.
  Arms: BioZ Group

SUMMARY:
Stroke volume variation (SVV) is an indicator used to assess the patient's volume status. The FloTrac system (Edwards Lifesciences, Irvine, CA) continuously monitors cardiac output (CO) and SVV (SVV-FloTrac) by analyzing the systemic arterial pressure wave. Numerous studies have demonstrated that SVV-FloTrac serves as a reliable indicator of fluid responsiveness. However, its peripheral invasiveness raises concerns about susceptibility to reflecting waves, damping, and vascular tone influences.In contrast, Transthoracic electrical bioimpedance (BioZ.com™) offers a non-invasive approach for continuously monitoring various hemodynamic variables. In this study, the primary aim was to assess the agreement between simultaneously measured SVV-FloTrac and SVV-BioZ.

ELIGIBILITY:
Inclusion Criteria:

* Age 18≤ Age ≤65
* patients undergoinglaparoscopic elective surgery for gastrointestinal tumors under general anesthesia
* 18 kg/m2≤BMI≤30 kg/m2
* ASA classification I-III
* Patients signed informed consent form

Exclusion Criteria:

* Arrhythmias
* The patient is diagnosed with severe cardiovascular disease（pulmonary arterial hypertension、left ventricular ejection fraction< 50%、aortic aneurysm、extensive peripheral arterial occlusive disease,、significant valvulopathy）
* Severe heart failure (METS<4)
* The patient is diagnosed with severe hepatic dysfunction (ChildePugh class C)
* The patient is diagnosed with severe renal dysfunction (undergoing dialysis before surgery)
* There is an infectious lesion on the skin or subcutaneous tissue where the non-invasive electrode piece is placed
* History of allergy to anesthetic drugs
* Weight<40kg
* Allergies to 6% hydroxyethyl starch, Fresenius Kabi, Deutschland

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The capacity to predict fluid responsiveness. | From anesthesia induction to the nonresponsive VLS about one hour.
  After anesthesia induction, volume loading was initiated. For each volume loading step (VLS), 100 mL of colloid solution (6% hydroxyethyl starch) was administered over a 2-minute duration. The SVV was measured and recorded simultaneously by FloTrac (SVV-FloTrac) and Transthoracic electrical bioimpedance(SVV-BioZ). Volume loading steps (VLS) continued until no responsive VLS was observed. Responsive VLS, defined as an increase in Flotrac-SV by at least 5%, and nonresponsive VLS, characterized by no change or an increase in Flotrac-SV by less than 5%, were subsequently identified. Multiple analysis methods were used to determine the capacity to predict the fluid responsiveness of these two devices.

SECONDARY OUTCOMES:
The agreement between simultaneously measured SVV-FloTrac and SVV-BioZ | From anesthesia induction to the nonresponsive VLS about one hour.
  After anesthesia induction, volume loading was initiated. For each volume loading step (VLS), 100 mL of colloid solution (6% hydroxyethyl starch) was administered over a 2-minute duration. The SVV was measured and recorded simultaneously by FloTrac (SVV-FloTrac) and Transthoracic electrical bioimpedance(SVV-BioZ). Volume loading steps (VLS) continued until no responsive VLS was observed. Responsive VLS, defined as an increase in Flotrac-SV by at least 5%, and nonresponsive VLS, characterized by no change or an increase in Flotrac-SV by less than 5%, were subsequently identified. Multiple analysis methods were used to determine the agreement of the two SVVs.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiaotong University School of Medicine, Pudong, Shanghai Municipality, China